CLINICAL TRIAL: NCT01027286
Title: Prospective Evaluation of Vitagel for Reduction in Blood Loss and Pain Following Unilateral Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Orthovita d/b/a Stryker (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-548
Record Dates: First submitted 2009-12-03; First posted 2009-12-07 (Estimated); Results first posted 2012-11-29 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-10

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitagel (Experimental)
  Interventions: Device: Vitagel
- Control (No Intervention): No Vitagel used.

INTERVENTIONS:
Device: Vitagel — Vitagel applied just prior to closure during primary total knee arthroplasty
  Arms: Vitagel

SUMMARY:
Vitagel® is an FDA approved class III medical device. It is a surgical hemostat, which has been shown to control bleeding during orthopaedic, cardiac, hepatic, and general surgical procedures. The product is a thrombin/collagen suspension which works in combination with the patient's own plasma to form a fibrin/collagen clot.

The present prospective, randomized controlled trial is designed to evaluate the efficacy of Vitagel® for reducing blood loss and pain in patients managed with unilateral total knee arthroplasty (TKA). It is hypothesized that the use of Vitagel® may lead to less blood filled knees, and thus to a greater improvement in postoperative pain scores when compared to the control group. The two arms of the study will include:

1. experimental group in which Vitagel® is used unilateral TKA
2. control group representing our current standard of care (no Vitagel®)

A comparison of the functional and clinical results between these two groups will be conducted using several outcome measures including the KOOS, SF-12 version2 and pain scores through the previously IRB approved OrthoMidas registry. The primary variable of interest is blood loss, based on hemoglobin drop during the postoperative hospital stay. Of secondary interest will be; 1) pain levels in the PACU, 2) pain scores for all postoperative days, 3) average pain for the entire hospital stay, 4) length of stay, 5) patient satisfaction at discharge, 4 weeks postoperative, and 12 weeks postoperative, and 6) functional scores at 4 and 12 weeks postoperative.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized, double-blinded, clinical trial involving three orthopaedic surgeons who perform total knee replacement. The proposed study is optimal for obtaining clinical and functional comparisons between TKA surgical procedures utilizing conventional practices (control) and TKA utilizing Vitagel®, a surgical hemostat used to control bleeding and facilitate healing. The study will include patients that are receiving a unilateral primary TKA.

Fifty cases will be assigned to each arm of the study (total 100 cases). This sample size was estimated using an alpha of 0.05 (conventional for all studies) and a beta of 0.80 (recommended for superiority studies). The standard deviation is based on a study conducted by the PI at the Cleveland Clinic in an IRB approved retrospective project in 2007, and will provide in excess of 80 percent statistical power in detecting less than a 100 ml difference in blood loss between the two groups.

The study will be conducted at the Cleveland Clinic (Cleveland, OH). The patients will not be informed of their treatment assignment, and the research investigator making observations and recording the data postoperatively will also be blinded to their treatment assignment. The placement of patients into treatment arms will be based on random drawing of sealed envelopes. An assessment of blinding will be conducted at the conclusion of the study by asking patients what treatment they think that they received.

Data will be collected at four timepoints, including preoperatively, during the hospital stay, 4 weeks postoperatively, and 12 weeks postoperatively. Preoperative data collected will include baseline SF-12, KOOS, hemoglobin and hematocrit levels, and pain scores. Data collected in the hospital will include hemoglobin and hematocrit levels, pain scores, narcotics usage, length of stay, and patient satisfaction at discharge. The SF-12, KOOS, pain scores, and patient satisfaction will be collected utilizing the 4 week (±2 weeks) standard of care postoperative visit. Patients are not always seen at the 12 week (±4 weeks) postoperative timepoint as standard of care. To collect these data, patients will be mailed the SF-12, KOOS, pain scores, patient satisfaction, and blinding assessment questionnaires. Patients not responding to the initial mailer will be contacted by phone and sent a second packet of questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 85 years
* Sex: Both male and female will be included. The male-to-female ratio will depend upon the patient population.
* Stable Health: At the time of surgery based on physical examination and medical history.
* Patient exhibited preoperative radiographic evidence of joint degeneration consistent with TKA that could not have been treated in non-operative fashion.
* Patient had severe knee pain and disability due to degenerative joint disease.
* Patient or patient's legal representative has signed the Informed Consent form. The patient is capable of making informed decisions regarding his/her healthcare.

Exclusion Criteria:

* Patients with history of liver disease. Patients with liver dysfunction from cirrhosis or hepatitis may have impaired production of factors in the clotting cascade which may make these individuals more prone to bleed, especially with the use of anticoagulants. For this reason, these patients will also be excluded from this study if a baseline INR if greater than 1.3.
* Patients allergic to materials of bovine origin.
* Patients predonating autologous blood.
* Patients with a preoperative platelet count of less than 100,000.
* Patients undergoing bilateral or revision surgery.
* Evidence of bleeding or metabolic - based hemolytic disorder (hemophilia or anticoagulation use), or hypercoaguable disorder.
* Previous history of infection in the affected joint.
* Peripheral vascular disease.
* Patient was a poor compliance risk - treated for ethanol or drug abuse, physical or mental handicap, etc.
* Patients with a previous history of venous thromboembolism, or other reason for requiring anticoagulation other than ASA 325 mg po BID and mechanical compression.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2009-07; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wael K Barsoum, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Result] Bloomfield MR, Klika AK, Molloy RM, Froimson MI, Krebs VE, Barsoum WK. Prospective randomized evaluation of a collagen/thrombin and autologous platelet hemostatic agent during total knee arthroplasty. J Arthroplasty. 2012 May;27(5):695-702. doi: 10.1016/j.arth.2011.09.014. Epub 2011 Oct 27. PMID 22035976

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitagel: Vitagel [Orthovita Inc., Malvern, PA], a collagen/thrombin and autologous platelet hemostatic agent, is applied just prior to surgical closure during primary total knee arthroplasty
- Control: No Vitagel used during primary total knee arthroplasty
Period: Overall Study
Arm/Group | Vitagel | Control
Started | 50 | 50
Preoperative | 50 | 50
Day of Surgery | 50 | 50
4 Week Postoperative | 49 | 50
12 Week Postoperative | 49 | 49
Completed | 49 | 49
Not Completed | 1 | 1
Not completed — Unable to Obtain Required Blood Volume | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitagel | Control | Total
Number analyzed (Participants) | 50 | 50 | 100
Age Continuous [Mean (Standard Deviation); unit: years] | 66.3 (8.2) | 62.4 (8.8) | 64.0 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 57
  Male | 22 | 21 | 43

OUTCOME MEASURES:

1. Secondary Outcome: Total Calculated Hospital Blood Loss
Time Frame: daily during hospital stay (an expected average of 4 days)
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Vitagel | Control
Number analyzed (Participants) | 49 | 50
mL | 1577 (541) | 1620 (565)

2. Primary Outcome: Number of Patients Managed With Blood Transfusion
Time Frame: daily during hospital stay (an expected average of 4 days)
Measure: Number; unit: participants
Arm/Group | Vitagel | Control
Number analyzed (Participants) | 49 | 50
participants | 0 | 5

3. Secondary Outcome: Preoperative & Postoperative Hemoglobin Values
Time Frame: within 30 days before surgery (preop), daily during hospital stay (an expected average of 4 days)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Vitagel | Control
Number analyzed (Participants) | 49 | 50
g/dL
  Preoperative | 13.8 (1.3) | 13.5 (1.4)
  Post Anesthesia Care Unit | 11.9 (1.3) | 11.8 (1.5)
  Postoperative Day 1 | 10.5 (1.2) | 10.4 (1.5)
  Postoperative Day 2 | 10.2 (1.2) | 9.7 (1.5)
  Postoperative Day 3 | 9.9 (1.3) | 9.4 (1.2)
  Postoperative Day 4 | 10.0 (1.0) | 8.8 (1.1)

4. Secondary Outcome: Daily Narcotic Usage (Morphine-equivalent mg)
Time Frame: daily during hospital stay (an expected average of 4 days)
Measure: Mean (Standard Deviation); unit: morphine-equivalent mg
Arm/Group | Vitagel | Control
Number analyzed (Participants) | 49 | 50
morphine-equivalent mg
  Postoperative Day 0 | 42.7 (35.0) | 50.5 (28.6)
  Postoperative Day 1 | 69.1 (49.7) | 74.8 (56.1)
  Postoperative Day 2 | 58.6 (47.2) | 65.4 (36.5)
  Postoperative Day 3 | 39.8 (42.2) | 52.3 (45.9)
  Postoperative Day 4 | 31.7 (43.2) | 45.8 (31.7)

5. Secondary Outcome: Length of Stay
Time Frame: day of hospital discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Vitagel | Control
Number analyzed (Participants) | 49 | 50
days | 3.3 (0.9) | 3.4 (0.8)

6. Secondary Outcome: Pain Score Scale
Description: A single scoring system used to evaluate overall pain on a scale of integers 0 to 10, with 0 representing "no pain" and 10 representing "unbearable pain." Thus, in this context, lower values represent better outcomes.
Time Frame: within 30 days before surgery (preop), 4 weeks after surgery, 12 weeks after surgery
Population: Vitagel (n=49 at preoperative, 4 wk, 12 wk); Control (n=50 at preoperative, 4 wk; n=49 at 12 wk since one control subject was lost to follow-up)
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Vitagel | Control
Number analyzed (Participants) | 49 | 50
points on a scale
  Preoperative | 5.5 (2.5) | 6.0 (2.4)
  4 Weeks Postoperative | 2.6 (2.1) | 2.5 (1.9)
  12 Weeks Postoperative | 1.9 (2.2) | 1.5 (1.4)

7. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: A scoring system used to evaluate the patient's opinion about his/her knee and associated problems. Subscales include 1) pain, 2) other symptoms, 3) function in daily living (ADL), 4) function in sport and recreation (Sport/Rec), and 5) knee related quality of life (QOL). Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score between 0 to 100 is calculated for each subscale. Subscale scores are generally not combined; rather, they are reported separated. Higher values represent better outcomes (i.e., less extreme symptoms).
Time Frame: within 30 days before surgery (preop), 4 weeks after surgery, 12 weeks after surgery
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Vitagel | Control
Number analyzed (Participants) | 49 | 50
points on a scale
  KOOS Pain: Preoperative | 43.5 (17.0) | 39.9 (16.8)
  KOOS Pain: 4 Wks Postoperative | 62.7 (20.4) | 57.1 (20.6)
  KOOS Pain: 12 Wks Postoperative | 76.6 (18.8) | 75.5 (14.6)
  KOOS Symptoms: Preoperative | 45.1 (18.6) | 39.6 (20.0)
  KOOS Symptoms: 4 Wks Postoperative | 61.9 (19.6) | 58.4 (16.8)
  KOOS Symptoms: 12 Wks Postoperative | 69.9 (19.2) | 68.5 (15.8)
  KOOS Daily Living Activities: Preoperative | 45.6 (20.9) | 45.8 (22.7)
  KOOS Daily Living Activities: 4 Wks Postoperative | 69.0 (19.5) | 67.7 (17.2)
  KOOS Daily Living Activities: 12 Wks Postoperative | 80.2 (16.5) | 81.2 (15.4)
  KOOS Sports/Recreation: Preoperative | 17.0 (22.6) | 12.2 (20.2)
  KOOS Sports/Recreation: 4 Wks Postoperative | 20.8 (29.2) | 28.1 (36.7)
  KOOS Sports/Recreation: 12 Wks Postoperative | 53.0 (31.8) | 51.6 (29.3)
  KOOS Quality of Life: Preoperative | 24.4 (24.3) | 27.7 (26.3)
  KOOS Quality of Life: 4 Wks Postoperative | 46.0 (29.0) | 51.0 (23.0)
  KOOS Quality of Life: 12 Wks Postoperative | 17.0 (22.6) | 12.2 (20.3)

ADVERSE EVENTS:
Arm/Group | Vitagel | Control
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 3/49 | 2/50
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitagel (N=49) | Control (N=50)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes